CLINICAL TRIAL: NCT04716803
Title: Bone Marrow Aspirate Concentrate (BMAC)Treatment for Knee Osteoarthritis
Acronym: BMAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kenneth Kalunian, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180916
Record Dates: First submitted 2020-11-03; First posted 2021-01-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Osteo Arthritis Knee
Keywords: moderate to severe knee osteoarthritis; total knee replacement; bone marrow; stem cell-based therapy; arthroscopy
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Bone marrow aspiration concentrate using the Angel System (Experimental): Bone marrow aspirate concentrate (BMAC) will be administered via injection to the knee of interest on day 14 of the study.
  Bone marrow aspiration will be concentrated using the Angel System.
  Interventions: Biological: Bone Marrow Aspirate Concentrate; Device: Angel Concentrated Platelet Rich Plasma (cPRP) System

INTERVENTIONS:
Biological: Bone Marrow Aspirate Concentrate — Aspiration of bone marrow will be collected from the patient's pelvic bone region and subsequently concentrated with the Angel Concentrated Platelet Rich Plasma (cPRP) System.
  Other Names: BMAC
Device: Angel Concentrated Platelet Rich Plasma (cPRP) System — Aspiration of bone marrow will be collected from the patient's pelvic bone region and subsequently concentrated with the Angel Concentrated Platelet Rich Plasma (cPRP) System.
  Other Names: The Angel System

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of bone marrow aspirate concentrate (BMAC) in patients with moderate to severe osteoarthritis of the knee. BMAC provides a rich source of mesenchymal stem cells (MSCs) and is a stem cell-based therapy that has been reported to preserve or improve the structure of joints. The Angel System is the device used in this study to concentrate bone marrow from the patient and is intended to separate a mixture of blood and bone marrow and collect plasma rich platelets preoperative to a surgical procedure. The goal of this study is to identify whether BMAC can be an effective and safe treatment for patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This is a pilot open-label, non-randomized, single institution study of BMAC administration in patient's with moderate to severe osteoarthritis of the knee who will undergo total knee replacement. Several weeks prior to total knee replacement, patients will have a sample of bone marrow taken from their pelvic region and concentrated using an investigational device called the Arthrex Angel Concentrated Platelet Rich Plasma (cPRP) System also known as the Angel System. The concentrated bone marrow will be immediately delivered back to the patient arthroscopically to the knee of interest. Blood and tissues samples will be collected at scheduled visits for molecular and histological analysis. Adverse events will be monitored throughout the trial. Assessment of healing will be performed by physical exam and standardized questionnaires related to the health of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Kellgren Lawrence radiographic grade IV
2. Need for a total knee arthroscopy by the patients primary care provider/or orthopedist.
3. Persistent pain in target knee that is unresponsive to standard of care including acetametaphine, non-steroidal anti-inflammatory drugs, physical therapy and/or intraarticular corticosteroids and/or hyaluronic acid preparations.
4. Males or females aged 45-75.

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients with at least one severe adverse event | End of Study (12 months)
  The number of life-threatening severe adverse events as determined by the standard FDA guidelines for adverse events that are deemed to be related to autologous BMAC concentrated by the Angel System and delivered via intra-articular injection into the knee.

SECONDARY OUTCOMES:
Structural change in knee from baseline measured by the VAS (Visual Analog Scale) in the American College of Rheumatology/Knee Osteoarthritis Assessment Scale (ACR/KOAS). | End of study (12 months)
  The VAS ranges from 0 to 100 with 0 indicating no damage and higher scores indicating more severe damage.
Self reported health from baseline through end of study measured by the 36-Item Short Form Survey Instrument (SF-36) Health Survey and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). | End of study (12 months)
  SF-36 scores are measured via ranges from 0 to 100.

OTHER OUTCOMES:
Rheumatic disease characterization | End of study (12 months)
  Biological samples (blood, urine, synovial tissue) are characterized via molecular and histological analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego Koman Outpatient Pavilion, La Jolla, California, United States